CLINICAL TRIAL: NCT07313839
Title: Comparison Between Double-Layer Self-Locking and Traditional Sutures in Post-Hysterectomy Laparoscopic Colporrhaphy: A Multicenter Pragmatic Randomized Controlled Trial
Brief Title: Comparison of Self-Locking Versus Traditional Sutures in Double-Layer Laparoscopic Vaginal Vault Closure After Hysterectomy (BI-SURE Trial)
Acronym: BI-SURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Vito Andrea Capozzi, Vito Andrea Capozzi, M.D. Department of Medicine and Surgery University Hospital of Parma, Parma, Italy, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 415/2024/DISP/AOUPR
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Gynecologic Cancers; Vaginal Cuff Dehiscence; Postoperative Complications
Keywords: Laparoscopic hysterectomy; Vaginal vault closure; Colporrhaphy; Self-locking suture; Barbed suture; Polyglactin 910; Gynecologic oncology; Postoperative complications; Randomized controlled trial
MeSH Terms: conditions — Postoperative Complications | interventions — Polyglactin 910

STUDY DESIGN:
Intervention Model Description: This is a multicenter, pragmatic, randomized controlled trial with a parallel assignment design. Eligible patients will be randomized in a 1:1 ratio to receive either double-layer self-locking sutures or double-layer traditional Polyglactin 910 sutures for laparoscopic vaginal vault closure following hysterectomy for gynecologic malignancy. The study is triple-blinded, with participants, outcome assessors, and statisticians masked to treatment allocation.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Self-Locking Suture Group (Experimental): Participants randomized to this arm will undergo laparoscopic vaginal vault closure after hysterectomy using a double-layer continuous suturing technique performed with a self-locking (barbed) suture, according to current clinical practice.
  Interventions: Procedure: Double-Layer Vaginal Vault Closure with Self-Locking Suture
- Traditional Suture Group (Active Comparator): Participants randomized to this arm will undergo laparoscopic vaginal vault closure after hysterectomy using a double-layer continuous suturing technique performed with traditional braided Polyglactin 910 suture, according to current clinical practice.
  Interventions: Procedure: Double-Layer Vaginal Vault Closure with Polyglactin 910

INTERVENTIONS:
Procedure: Double-Layer Vaginal Vault Closure with Self-Locking Suture — Laparoscopic vaginal vault closure performed using a double-layer continuous suturing technique with a self-locking (barbed) suture following hysterectomy.
  Arms: Self-Locking Suture Group
Procedure: Double-Layer Vaginal Vault Closure with Polyglactin 910 — Laparoscopic vaginal vault closure performed using a double-layer continuous suturing technique with traditional braided Polyglactin 910 suture following hysterectomy.
  Arms: Traditional Suture Group

SUMMARY:
Vaginal vault closure after laparoscopic or robotic hysterectomy may be associated with postoperative complications such as vaginal cuff dehiscence, infection, and bleeding. The optimal suture material and technique for laparoscopic colporrhaphy, particularly in patients undergoing surgery for gynecologic malignancies, remain controversial.

The BI-SURE trial is a multicenter, randomized controlled study designed to compare double-layer self-locking sutures versus double-layer traditional Polyglactin 910 sutures for laparoscopic vaginal vault closure after hysterectomy. The study aims to evaluate postoperative effectiveness and safety within three months after surgery.

DETAILED DESCRIPTION:
Laparoscopic and robotic hysterectomy represent standard surgical approaches for the treatment of gynecologic malignancies but are associated with a higher risk of vaginal vault complications compared with open or vaginal surgery. Although uncommon, postoperative complications such as vaginal cuff dehiscence, infection, and bleeding may lead to significant morbidity and require additional medical or surgical interventions.

Vaginal vault closure can be performed using different suturing techniques and materials. Traditional braided sutures, such as Polyglactin 910, are widely used in clinical practice, while self-locking (barbed) sutures have been introduced to facilitate laparoscopic suturing by maintaining tissue approximation without the need for knots. Evidence comparing these sutures is limited, particularly for double-layer closure techniques and in patients treated for gynecologic malignancies.

The BI-SURE trial is a multicenter, pragmatic, randomized controlled trial designed to compare double-layer self-locking sutures versus double-layer traditional Polyglactin 910 sutures for laparoscopic vaginal vault closure following hysterectomy for malignant gynecologic disease. Eligible patients will be randomized in a 1:1 ratio. Postoperative outcomes will be assessed up to three months after surgery, including vaginal cuff-related complications and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic or robotically assisted hysterectomy for gynecologic malignant disease
* Age ≥ 18 years
* Ability to provide written informed consent

Exclusion Criteria:

* Laparotomic or vaginal hysterectomy
* Contraindication to laparoscopic vaginal vault closure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal cuff dehiscence rate | Within 3 months after surgery
  Proportion of participants experiencing vaginal cuff dehiscence requiring surgical reintervention after laparoscopic hysterectomy.
Vaginal cuff infection rate | Within 3 months after surgery
  Proportion of participants developing vaginal cuff infection, defined as abnormal vaginal discharge with or without fever, leukocytosis, and/or local tenderness, requiring antibiotic therapy.
Postoperative bleeding rate | Within 3 months after surgery
  Proportion of participants experiencing postoperative vaginal cuff bleeding requiring hemostatic treatment.

SECONDARY OUTCOMES:
Postoperative pain intensity | At 1 month and 3 months after surgery
  Postoperative pain assessed using the Visual Analogue Scale (VAS).
Early postoperative composite complication rate | Within 1 month after surgery
  Proportion of participants experiencing vaginal cuff dehiscence, infection, or bleeding before the initiation of adjuvant therapy.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Department of Medicine and Surgery, University Hospital of Parma, Parma, Italy
  - Division of Oncologic Gynecology, IRCCS Azienda Ospedaliero-Universitaria di Bologna, 40138 Bologna, Italy., Bologna
  - Department of Obstetrics and Gynecology, Ospedale Santa Croce e Carle, Cuneo, Italy., Cuneo
  - Department of Gynecologic Oncology. Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Italy., Milan
  - Clinic of Obstetrics and Gynecology, "Santa Maria della Misericordia" University Hospital, Azienda Sanitaria Universitaria Friuli Centrale, Udine, Italy., Udine

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is conducted within a hospital-based academic setting and no data repository has been designated for public data release. Data will be stored securely at the sponsor institution and will be accessible only to authorized study personnel in compliance with applicable privacy regulations.